CLINICAL TRIAL: NCT06754384
Title: Randomized, Double-blind, Controlled Phase I/II Clinical Trial on the Tolerability, Safety, and Immunogenicity of Tetravalent Inactivated Enterovirus Vaccine (Vero Cell) in Healthy Adults and Children Aged 6 Months to 12 Years.
Brief Title: Tolerability, Safety, and Immunogenicity of Tetravalent Inactivated Enterovirus Vaccine (Vero Cell).
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-QEV-1001
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Hand, Foot, and Mouth Disease (HFMD); Herpangina
Keywords: Phase Ⅰ; phase Ⅱ; tolerability; safety; immunogenicity; Hand, Foot, and Mouth Disease (HFMD); Herpangina
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Herpangina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-dose of tetravalent inactivated enterovirus vaccine (Vero cell) (Experimental): Low-dose of tetravalent inactivated enterovirus vaccine (Vero cell)(Only for phase Ⅰ)
  Interventions: Biological: Low-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
- Medium-dose of tetravalent inactivated enterovirus vaccine (Vero cell) (Experimental): Medium-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
  Interventions: Biological: Medium-dose tetravalent inactivated enterovirus vaccine (Vero cell)
- High-dose of tetravalent inactivated enterovirus vaccine (Vero cell) (Experimental): High-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
  Interventions: Biological: High-dose tetravalent inactivated enterovirus vaccine (Vero cell) )
- EV71 vaccine (Active Comparator): EV71 vaccine (for ages 6-71 months)
  Interventions: Biological: EV71 inactivated enterovirus vaccine (Vero cell) )(for ages 6-71 months）
- placebo (Placebo Comparator): placebo (for ages 6-12 years)
  Interventions: Biological: placebo (for ages 6-12 years)

INTERVENTIONS:
Biological: Low-dose of tetravalent inactivated enterovirus vaccine (Vero cell) — Low-dose tetravalent inactivated enterovirus vaccine (Vero cell) )(only for phase Ⅰ）
  Arms: Low-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
Biological: Medium-dose tetravalent inactivated enterovirus vaccine (Vero cell) — Medium-dose tetravalent inactivated enterovirus vaccine (Vero cell)
  Arms: Medium-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
Biological: High-dose tetravalent inactivated enterovirus vaccine (Vero cell) ) — High-dose tetravalent inactivated enterovirus vaccine (Vero cell) )
  Arms: High-dose of tetravalent inactivated enterovirus vaccine (Vero cell)
Biological: EV71 inactivated enterovirus vaccine (Vero cell) )(for ages 6-71 months） — EV71 inactivated enterovirus vaccine (Vero cell) )(for ages 6-71 months）
  Arms: EV71 vaccine
Biological: placebo (for ages 6-12 years) — placebo (for ages 6-12 years)
  Arms: placebo

SUMMARY:
The trial aims to assess the tolerability, safety, and immunogenicity of the tetravalent inactivated enterovirus vaccine in adults and children aged 6 months to 12 years. The main questions it aims to answer are:

* Phase Ⅰ: The safety of the investigational vaccine in the target population based on adverse events (AEs);
* Phase Ⅱ: The immunogenicity of the investigational vaccine in the target population.

In Phase I, researchers will compare the safety of the investigational vaccine at low, medium, and high doses with the control vaccine; in Phase II, they will compare the safety and immunogenicity (including immune persistence) of the investigational vaccine at medium and high doses with the control vaccine.

Procedure:

* In Phase I, will be vaccinated with the investigational vaccine (at low, medium, and high doses) or the control EV71 vaccine/placebo in a 3:1 ratio, following a vaccination schedule of 0 and 1 month. Within each age group, and under the premise of ensuring safety, a dose-escalation trial will be conducted in reverse order of age.
* In Phase II, participants in each age group will be randomly assigned to the medium-dose, high-dose investigational vaccine groups, and the control group in a 1:1:1 ratio, receiving two doses of the investigational vaccine or the EV71 vaccine (for ages 6-71 months)/placebo (for ages 6-12 years), with a one-month interval between the two doses.
* For all participants in both Phase I and Phase II, immediate reactions within 30 minutes after each dose will be observed. Diary cards/contact cards will be used to collect solicited local and systemic adverse events (AEs) for 0-7 days and unsolicited AEs for 0-30 days after vaccination. Additionally, serious adverse events (SAEs) will be monitored from the start of vaccination until 6 months post-completion of the vaccination schedule. Furthermore, for participants of reproductive age in Phase I, pregnancy events will be collected.

DETAILED DESCRIPTION:
Both Phase I and Phase II clinical trials adopt a randomized, double-blind, controlled design.

For Phase I, 192 healthy participants are planned to be enrolled, including 48 adults aged 18-59, 48 children aged 6-12, 48 children aged 24-71 months, and 48 children aged 6-23 months. They will receive two doses of the experimental vaccine or EV71 vaccine (for those aged 6-71 months) / placebo (for those aged 6-12 and 18-59) in the order of low-dose, medium-dose, and high-dose. The interval between the two doses is one month. Enrollment will follow the sequence of adults aged 18-59, children aged 6-12, children aged 24-71 months, and children aged 6-23 months. Within each dosage stage, there will be 16 participants from each age group, and they will receive the experimental vaccine or control EV71 vaccine / placebo in a 3:1 ratio.

The dose escalation principle within each age group is low-dose, medium-dose, and high-dose. Based on the occurrence of AEs and clinical laboratory indicators, the next higher dose stage can only be initiated after a 0-7 day safety observation period following the first dose of the lower dose stage and confirmation of safety. The sequential enrollment principle across age groups is adults aged 18-59, children aged 6-12, children aged 24-71 months, and children aged 6-23 months. For each dose, after completing the 0-7 day safety observation period following the first dose and confirming safety, the next age group can proceed with enrollment for that dose.

For adults aged 18-59 and children aged 6-12, venous blood and urine samples will be collected before each dose and on the 3rd day after vaccination for blood routine tests (about 2.0 ml of venous blood), blood biochemistry tests (about 2.0-3.0 ml of venous blood), and urine routine tests (about 2.0-10.0 ml of urine) to evaluate vaccine safety. For children aged 24-71 months, only about 2.0-3.0 ml of venous blood will be collected at the corresponding time points for blood biochemistry tests.

If more than 10% of participants in each dose stage of the 24-71 month age group experience abnormal laboratory test results related to the investigational vaccine and of clinical significance after the first dose, then for the corresponding dose stage in the 6-23 month age group, blood routine tests (about 1.0 ml of venous blood), blood biochemistry tests (about 2.0-3.0 ml of venous blood), and urine routine tests (about 2.0-10.0 ml of urine) will be conducted on the 3rd day after the first dose, before the second dose, and on the 3rd day after the second dose.

After obtaining safety data for all participants in Phase I for 30 days after the completion of vaccination, the data will be analyzed, and a safety analysis report will be submitted to the Data Monitoring Committee (DMC) and Ethical Committee (EC) for review. Only after confirming safety can the Phase II clinical trial be initiated.

For Phase II, 360 healthy participants aged 6 months to 12 years are planned to be enrolled, including 120 children aged 6-23 months, 120 children aged 24-71 months, and 120 children aged 6-12. Participants in each age group will be randomly assigned to the medium-dose and high-dose groups of the investigational vaccine and the control group in a 1:1:1 ratio, receiving two doses of the investigational vaccine or EV71 vaccine (for those aged 6-71 months) / placebo (for those aged 6-12) with a one-month interval. With the day of the first dose as Day 0, all participants in Phase II will have about 3.0 ml of venous blood collected on Days 0, 60, and 210 to separate serum for EV71, CA16, CA10, and CA6 neutralizing antibody tests, evaluating the vaccine's immunogenicity and immune persistence.

All participants in both Phase I and Phase II will be observed for immediate reactions within 30 minutes after each dose, and solicited local and systemic AEs will be collected for 0-7 days, while unsolicited AEs will be collected for 0-30 days. Additionally, SAE monitoring will be conducted from the start of vaccination until 6 months after the completion of the vaccination schedule. Furthermore, for fertile participants in the Phase I clinical trial, during the trial and after the first dose, pregnancy events of female participants themselves or the partners of male participants will be collected through a combination of active follow-up by researchers and self-reporting by participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18-59 years (only applicable for Phase I) or 6 months to 12 years.
* Participants and/or their legal guardians are able to understand and voluntarily sign the informed consent form (for participants aged 8-12, both the participant and their guardian must sign).
* Willing and able to comply with all visit schedules, sample collection, vaccinations, and other trial procedures, and maintain contact during the trial period.
* Provide identification for the participant and/or their guardian.
* Participants of childbearing participants and their sexual partners must voluntarily use effective contraceptive measures from the time of signing the informed consent form until three months after the completion of the two-dose vaccination series with the investigational vaccine, and have no plans to donate sperm or ova (only applicable for Phase I participants aged 18-59 years).

Exclusion Criteria:

* History of HFMD or HA (only applicable to Phase II clinical trial participants).
* Presence of uncontrolled chronic diseases or history of serious illnesses, including but not limited to cardiovascular diseases, hematological diseases, liver and kidney diseases, digestive system diseases, respiratory diseases, malignant tumors, and history of major organ transplantation.
* Severe congenital malformations, genetic defects, or malnutrition.
* Presence of autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, asplenia, functional asplenia, HIV infection).
* Abnormal coagulation function (such as coagulation factor deficiency, platelet abnormalities).
* Suffering from/having suffered from severe neurological diseases (epilepsy, convulsions, or seizures [excluding febrile convulsions]), mental illness, or having a family history of mental illness.
* Acute illnesses or acute exacerbations of chronic illnesses within the past 3 days.
* Having been vaccinated with a vaccine containing any of the components EV71, CA16, CA10, CA6 (including marketed vaccines or investigational vaccines).
* Having received ≥14 days of immunosuppressive or other immunomodulatory treatment (adults: prednisone ≥20mg/day, or children: ≥2mg/kg/day, or equivalent doses; excluding topical or inhaled corticosteroids) within the past 6 months, or cytotoxic treatment, or planning to receive such treatment during the trial.
* Having received immunoglobulins or other blood products within the past 6 months, or planning to receive such treatment during the trial.
* Having received other investigational drugs or vaccines within the past 30 days, or planning to receive such drugs or vaccines during the trial.
* Having received live attenuated vaccines or nucleic acid vaccines within the past 14 days, or subunit or inactivated vaccines within the past 7 days.
* Known allergy to any component of the investigational vaccine (inactivated EV71, CA16, CA10, and CA6 viruses, aluminum hydroxide adjuvant, disodium phosphate, sodium dihydrogen phosphate, sodium chloride, water for injection).
* Participants who are breastfeeding, pregnant, or planning to become pregnant within 3 months after the two doses of vaccination in this trial (only applicable to Phase I).
* On the day of planned vaccination with the investigational vaccine, having an axillary temperature >37.0°C before vaccination, or other vital sign measurements outside the normal range.
* Failing the physical examination on the day of planned vaccination with the investigational vaccine.
* Clinically significant laboratory abnormalities beyond the reference range in clinical laboratory tests (only applicable to Phase I clinical trial participants):

  1. Hematology-related test indicators (adults aged 18-59 and children aged 6- white blood cell count, hemoglobin, and platelet count.
  2. Blood chemistry-related test indicators (adults aged 18-59, children aged 6-12, and children aged 24-71 months): alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), fasting blood glucose.
  3. Urinalysis-related test indicators (adults aged 18-59 and children aged 6-12): urine protein (PRO).
* Presence of skin lesions, inflammation, ulcers, rashes, scars, or other conditions at the intended injection site that may interfere with vaccination or observation of local reactions.
* Any other factors deemed by the investigator to make the participant unsuitable for participation in the clinical trial.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 552 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ⅰ:The safety of the investigational vaccine in the target population based on AR. | 60 days
  Incidence rate of AR from vaccination onset to 30 days post-full immunization in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate the seropositive conversion rates of the investigational vaccine in the target population. | 60 days
  The seropositive conversion rates of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate the geometric mean titer (GMT) of the investigational vaccine in the target population. | 60 days
  The GMT of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 months to 12 years.

SECONDARY OUTCOMES:
phase Ⅰ:Evaluate the safety of the investigational vaccine in the target population based on adverse events (AEs). | 60 days
  Incidence rate of adverse reactions (ARs) from vaccination onset to 30 days post full immunization in adults aged 18-59.
phase Ⅰ: Evaluate the safety of the investigational vaccine in the target population based on adverse events (AEs) in adults aged 18-59. | 7 monthes
  phase Ⅰ: Incidence rate of serious adverse events (SAEs) from vaccination onset to 6 months post full immunization in adults aged 18-59.
phase Ⅰ: Evaluate the safety of the investigational vaccine in the target population based on AEs in children aged 6 months to 12 years. | 7 monthes
  phase Ⅰ: Incidence rate of serious adverse events (SAEs) from vaccination onset to 6 months post full immunization in children aged 6 months to 12 years.
phase Ⅰ:Evaluate the safety of the investigational vaccine in adults aged 18-59 and children aged 6-12 based on laboratory abnormalities. | 3 days
  Incidence rate of clinically significant abnormalities in blood biochemistry, blood routine, and urinalysis indicators on the 3rd day after each dose in adults aged 18-59 and children aged 6-12.
phase Ⅰ:Evaluate the safety of the investigational vaccine in children aged 24-71 months based on laboratory abnormalities. | 3 days
  phase Ⅰ:Incidence rate of clinically significant abnormalities in blood biochemistry indicators on the 3rd day after each dose in children aged 24-71 months.
phase Ⅱ:Evaluate the seropositive rate of the investigational vaccine. | 60 days
  phase Ⅱ: Seropositive rate and of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate Geometric mean increase (GMI) of the investigational vaccine in children aged 6 months to 12 years. | 60 days
  Phase Ⅱ: GMI of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate the seroconversion rate of the investigational vaccine in children aged 6 to 71 months. | 60 days
  Phase Ⅱ:Seroconversion rate of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 71 months.
Phase Ⅱ:Evaluate the seropositive rate of the investigational vaccine in children aged 6 to 71 months. | 60 days
  Phase Ⅱ:Seropositive rate of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 71 months.
Phase Ⅱ:Evaluate the GMT of the investigational vaccine in children aged 6 to 71 months. | 60 days
  Phase Ⅱ: GMT of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 71 months.
Phase Ⅱ:Evaluate the GMI of the investigational vaccine in children aged 6 to 71 months. | 60 days
  Phase Ⅱ: GMI of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 71 months.
Phase Ⅱ:Evaluate the seroconversion rate of the investigational vaccine in children aged 6 to 12 years. | 60 days
  Phase Ⅱ:Seroconversion rate of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 12 years.
Phase Ⅱ:Evaluate the seropositive rate of the investigational vaccine in children aged 6 to 12 years | 60 days
  Phase Ⅱ:Seropositive rate of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 12 years.
Phase Ⅱ:Evaluate the GMT of the investigational vaccine in children aged 6 to 12 years. | 60 days
  Phase Ⅱ: GMT of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 12 years.
Phase Ⅱ:Evaluate the GMI of the investigational vaccine in children aged 6 to 12 years. | 60 days
  Phase Ⅱ: GMI of neutralizing antibodies against EV71, CA16, CA10, and CA6 on the 30th day after full vaccination in children aged 6 to 12 years.
phase Ⅱ:Evaluate the safety of the investigational vaccine based on AEs. | 60 days
  phase Ⅱ:Incidence rate of ARs from vaccination onset to 30 days post full immunization in children aged 6 months to 12 years.
phase Ⅱ:Evaluate the safety of the investigational vaccine based on AEs. | 7 monthes
  phase Ⅱ:Incidence rate of SAEs from vaccination onset to 6 months post full immunization in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate the immune persistence of the investigational vaccine via seropositive rate of neutralizing antibodies. | 7 monthes
  Phase Ⅱ: Seropositive rate of neutralizing antibodies against EV71, CA16, CA10, and CA6 at 6 months post full immunization in children aged 6 months to 12 years.
Phase Ⅱ:Evaluate the immune persistence of the investigational vaccine via GMT of neutralizing antibodies. | 7 monthes
  Phase Ⅱ: GMT of neutralizing antibodies against EV71, CA16, CA10, and CA6 at 6 months post full immunization in children aged 6 months to 12 years.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shenyu, Dr., Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided